CLINICAL TRIAL: NCT04931680
Title: Risk Factors for Treatment Failure of Scabies in Autochthonous Populations of French Guiana (GUYAGALE)
Acronym: GUYAGALE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: GUYAGALE
Record Dates: First submitted 2021-05-11; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Scabies
Keywords: Scabies; Risk Factors; Prevalence; Indigenous Population
MeSH Terms: conditions — Scabies | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with treatment success: Patients with diagnosis of "confirmed" or "clinical" scabies and treatment success
  Interventions: Other: Data collection
- Patients with treatment failure: Patients with diagnosis of "confirmed" or "clinical" scabies and treatment failure
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — During the follow-up consultation, six weeks after inclusion (S6), data will be collected using a standardized digital questionnaire, including clinical features, economic, social and cultural characteristics, housing conditions and therapeutic details (type of environmental decontamination and treatment received). Data will then be compared between patients with therapeutic success or failure. A urine test strip will also be used during the S6 consultation to screen for proteinuria. The prevalence of post-streptococcal glomerulonephritis will be extrapolated from that of proteinuria.

SUMMARY:
Scabies is a Neglected Tropical Disease, particularly important in autochthonous populations. Treatment failures could explain the high prevalence of this disease in Amerindian and Maroon populations of French Guiana. Our main objective is to look for specific sociodemographic risk factors for treatment failure of scabies in the remote areas of French Guiana. A secondary objective is to evaluate the prevalence of scabies and its complications.

DETAILED DESCRIPTION:
Scabies is known to be a health issue of particular importance in marginal and autochthonous populations throughout the world. French Guiana is a French territory harbouring several autochthonous populations living in remote rainforest areas. The prevalence of scabies remains high in these areas despite primary care offered by the local health centres. A prevalence of 2.5% was found in two Amerindian villages in a retrospective study in 2019. Therapeutic failures are known to be one of the main causes of a long-lasting high prevalence. In low-resources populations, socio-economic factors and promiscuity are particularly incriminated. The role played by these factors should be studied in French Guiana. Secondary complications such as impetigo and post-streptococcal glomerulonephritis should be evaluated, as they represent an important part of the global burden of scabies.

This study will be conducted from April to August 2021 in remote settlements of French Guiana. Patients will be seen during a first inclusion consultation, realized by the same investigator (RB). All patients with diagnosis of " confirmed " or " clinical " scabies according to the International Alliance for the Control of Scabies will be included in case of agreement. Patients will be treated according to the current protocol in the Health Centres for Remote Areas of French Guiana (according to the European guidelines for the treatment of scabies: two doses of ivermectin 0.2mg/kg on day 1 and day 7 ; benzyl benzoate 10% or permethrin 5% for children under 15kg or pregnant women). The follow-up consultation will take place six weeks later. The same investigator (RB) will assess treatment failure or success.

Research of etiologic factors associated with treatment failure; multicentric regional sample

Category 3 Non-Interventional Human Person Research (RIPH 3)

ELIGIBILITY:
* Inclusion criteria :

  * Confirmed or clinical scabies according to the criteria of the International Alliance for the Control of Scabies
  * Agreement to answer to the follow-up questionnaire
  * Agreement to come back for a six-weeks follow-up consultation.
* Exclusion criteria:

  * Patient with possible diagnosis of scabies, not fulfilling the criteria for " confirmed " or " clinical " scabies
  * Refusal of the questionnaire or the follow-up consultation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with diagnosis of " confirmed " or " clinical " scabies according to the International Alliance for the Control of Scabies will be included in case of agreement.
Sampling Method: Non-Probability Sample
Enrollment: 276 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-25 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment failure of scabies | Six weeks after enrollment (S6)
  Number of participants with treatment failure of scabies (persistance of cutaneous lesions), six weeks after enrollment (S6)

SECONDARY OUTCOMES:
Confirmed or clinical diagnosis of scabies | At enrollment (D0) - one day
  Confirmed or clinical diagnosis of scabies : at enrollment (D0)
Presence of impetigo | At enrollment (D0) - one day
  Presence of impetigo : at enrollment (D0)
Presence of proteinuria | Six weeks after enrollment (S6)
  Presence of proteinuria : six weeks after enrollment (S6)

OTHER OUTCOMES:
Qualitative study by semi-structured questionnaire | Six weeks after enrollment (S6)
  Qualitative study by questionnaire performed by a trained anthropologist to determine the knowledge, attitudes and practices of patients infected with scabies in the study area (S6)

CONTACTS AND LOCATIONS:
Overall Officials: Romain BLAIZOT, MD, Principal Investigator — Centre Hospitalier de Cayenne
Locations (1):
- General Hospital of Cayenne, Cayenne, French Guiana

REFERENCES:
- [Background] Engelman D, Cantey PT, Marks M, Solomon AW, Chang AY, Chosidow O, Enbiale W, Engels D, Hay RJ, Hendrickx D, Hotez PJ, Kaldor JM, Kama M, Mackenzie CD, McCarthy JS, Martin DL, Mengistu B, Maurer T, Negussu N, Romani L, Sokana O, Whitfeld MJ, Fuller LC, Steer AC. The public health control of scabies: priorities for research and action. Lancet. 2019 Jul 6;394(10192):81-92. doi: 10.1016/S0140-6736(19)31136-5. Epub 2019 Jun 6. PMID 31178154